CLINICAL TRIAL: NCT05307471
Title: Physiopathologic Study of Induced by Thoracotomy / Thoracoscopy Neuropathy Mechanism Clinical, Psychophysical, Electrophysiological Approach, and in Response to Therapy
Brief Title: Physiopathologic Study of Induced by Thoracotomy / Thoracoscopy Neuropathy Mechanism
Acronym: NITT
Status: Terminated | Type: Observational
Why Stopped: No neuropathic pain in recruited subjects
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0161; 2012-A00905-38 (Other: IDRCB)
Record Dates: First submitted 2013-06-25; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2021-11

CONDITIONS: Thoracotomy; Thoracoscopy
Keywords: Thoracotomy; Thoracoscopy; Neuropathy; Neuropathic pain; Pulmonary surgery
MeSH Terms: conditions — Neuralgia | interventions — Thoracotomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- neuropathic pain: This study will be proposed to patients undergoing thoracotomy or thoracoscopy for partial or total lung resection in the service of Thoracic Surgery of Centre Jean Perrin (Prof. M. Filaire), the objective is to recruit 120 patients (for 100 evaluable patients) over a period of 18 months of inclusion
  Interventions: Other: Thoracotomy/scopy

INTERVENTIONS:
Other: Thoracotomy/scopy

SUMMARY:
Pulmonary surgery, performed routinely by thoracotomy or thoracoscopy, can cause significant and frequent chronic postoperative pain, most often neuropathic. The role of trauma intraoperative intercostal nerve is evoked to explain the genesis of the neuropathy. Treatments proposed in the indication of neuropathic pain in a broad sense, are exposed to many cases of failures. It is supposed that these failures are due to a mismatch between the selected drug (which is specific to the target) and the real pathology because neuropathy encompasses many different pathophysiological syndromes which are sometimes intricated.

The main objective of this project is to study the clinical, psychophysical and electrophysiological (noninvasively) intercostal nerve affected by the surgery at the second postoperative month, by comparing the results with similar observations made shortly before the intervention.

This study will be proposed to patients undergoing thoracotomy or thoracoscopy for partial or total lung resection in the service of Thoracic Surgery of Centre Jean Perrin, the objective is to recruit 120 patients (for 100 evaluable patients) over a period of 18 months of inclusion.

The other objective of the project is to provide a treatment algorithm for patients in pain, and to compare the efficacy of this treatment with the pre-treatment observations data.

DETAILED DESCRIPTION:
Exploratory study, including additional examinations and visits. Biomedical research.

ELIGIBILITY:
Inclusion criteria :

* patients undergoing lateral or posterolateral thoracotomy scheduled lung surgery, regardless of indication, or lung or pleural scheduled surgery (treatment of recurrent pneumothorax) by thoracoscopy;
* 18 to 80 years
* Informed consent to the trial
* Protected by the French health welfare

Exclusion Criteria:

* Refusal of the patient;
* Preexisting neuropathy ;
* Treatment of active substance known on neuropathic pain: gabapentin, pregabalin, amitryptyline, duloxetine, venlafaxine, tricyclic antidepressants, topical lidocaine or capsaicin;
* Emergency surgery;
* Specific clinical contexts including terminal or palliative neoplasia;
* Deficit psychiatric pathology and dementia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing thoracotomy or thoracoscopy for partial or total lung resection
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2013-10-28 (Actual); Primary Completion 2017-04-12 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Presence of spontaneous pain on the operated hemithorax | Day 0 (day of surgery)
  Patient interview (yes/no)
Presence of spontaneous pain on the operated hemithorax | Visit 2 = 2 months after Day 0 (day of surgery)
  Patient interview (yes/no)
Presence of spontaneous pain on the unoperated hemithorax | Day 0 (day of surgery)
  Patient interview (yes/no)
Presence of spontaneous pain on the unoperated hemithorax | Visit 2 = 2 months after Day 0 (day of surgery)
  Patient interview (yes/no)
Intensity of spontaneous pain on the operated hemithorax | Day 0 (day of surgery)
  Numeric scale of value (from 0 to 10)
Intensity of spontaneous pain on the operated hemithorax | Visit 2 = 2 months after Day 0 (day of surgery)
  Numeric scale of value (from 0 to 10)
Intensity of spontaneous pain on the unoperated hemithorax | Day 0 (day of surgery)
  Numeric scale of value (from 0 to 10)
Intensity of spontaneous pain on the unoperated hemithorax | Visit 2 = 2 months after Day 0 (day of surgery)
  Numeric scale of value (from 0 to 10)
Characteristics of spontaneous pain on the operated hemithorax | Day 0 (day of surgery)
  Neuropathic Pain Symptom Inventory (NPSI) survey
Characteristics of spontaneous pain on the operated hemithorax | Visit 2 = 2 months after Day 0 (day of surgery)
  Neuropathic Pain Symptom Inventory (NPSI) survey
Characteristics of spontaneous pain on the unoperated hemithorax | Day 0 (day of surgery)
  Neuropathic Pain Symptom Inventory (NPSI) survey
Characteristics of spontaneous pain on the unoperated hemithorax | Visit 2 = 2 months after Day 0 (day of surgery)
  Neuropathic Pain Symptom Inventory (NPSI) survey
Measurement of threshold sensitivity to cold on the operated hemithorax | Day 0 (day of surgery)
  The thermode will be applied and patients will be asked to press a button when a cold sensation will be first perceived, thus defining the thermal threshold for that stimulus presentation.
Measurement of threshold sensitivity to cold on the operated hemithorax | Visit 2 = 2 months after Day 0 (day of surgery)
  The thermode will be applied and patients will be asked to press a button when a cold sensation will be first perceived, thus defining the thermal threshold for that stimulus presentation.
Measurement of threshold sensitivity to cold on the unoperated hemithorax | Visit 2 = 2 months after Day 0 (day of surgery)
  The thermode will be applied and patients will be asked to press a button when a cold sensation will be first perceived, thus defining the thermal threshold for that stimulus presentation.
Measurement of threshold sensitivity to hot on the operated hemithorax | Day 0 (day of surgery)
  The thermode will be applied and patients will be asked to press a button when a hot sensation will be first perceived, thus defining the thermal threshold for that stimulus presentation.
Measurement of threshold sensitivity to hot on the operated hemithorax | Visit 2 = 2 months after Day 0 (day of surgery)
  The thermode will be applied and patients will be asked to press a button when a hot sensation will be first perceived, thus defining the thermal threshold for that stimulus presentation.
Measurement of threshold sensitivity to hot on the unoperated hemithorax | Visit 2 = 2 months after Day 0 (day of surgery)
  The thermode will be applied and patients will be asked to press a button when a hot sensation will be first perceived, thus defining the thermal threshold for that stimulus presentation.
Measurement of nociceptive threshold sensitivity to cold on the operated hemithorax | Day 0 (day of surgery)
  The thermode will be applied and patients will be asked to press a button when a cold painful sensation will be first perceived, thus defining the thermal nociceptive threshold for that stimulus presentation.
Measurement of nociceptive threshold sensitivity to cold on the operated hemithorax | Visit 2 = 2 months after Day 0 (day of surgery)
  The thermode will be applied and patients will be asked to press a button when a cold painful sensation will be first perceived, thus defining the thermal nociceptive threshold for that stimulus presentation.
Measurement of nociceptive threshold sensitivity to cold on the unoperated hemithorax | Visit 2 = 2 months after Day 0 (day of surgery)
  The thermode will be applied and patients will be asked to press a button when a cold painful sensation will be first perceived, thus defining the thermal nociceptive threshold for that stimulus presentation.
Measurement of nociceptive threshold sensitivity to hot on the operated hemithorax | Day 0 (day of surgery)
  The thermode will be applied and patients will be asked to press a button when a hot painful sensation will be first perceived, thus defining the thermal nociceptive threshold for that stimulus presentation.
Measurement of nociceptive threshold sensitivity to hot on the operated hemithorax | Visit 2 = 2 months after Day 0 (day of surgery)
  The thermode will be applied and patients will be asked to press a button when a hot painful sensation will be first perceived, thus defining the thermal nociceptive threshold for that stimulus presentation.
Measurement of nociceptive threshold sensitivity to hot on the unoperated hemithorax | Visit 2 = 2 months after Day 0 (day of surgery)
  The thermode will be applied and patients will be asked to press a button when a hot painful sensation will be first perceived, thus defining the thermal nociceptive threshold for that stimulus presentation.
Measurement of threshold tactile sensitivity on the operated hemithorax | Day 0 (day of surgery)
  Thickness of the 1st filament felt by the patient by application of Von Frey filaments of increasing size from 0.008 to 300 grams in pressure equivalent
Measurement of threshold tactile sensitivity on the operated hemithorax | Visit 2 = 2 months after Day 0 (day of surgery)
  Thickness of the 1st filament felt by the patient by application of Von Frey filaments of increasing size from 0.008 to 300 grams in pressure equivalent
Measurement of threshold tactile sensitivity on the unoperated hemithorax | Visit 2 = 2 months after Day 0 (day of surgery)
  Thickness of the 1st filament felt by the patient by application of Von Frey filaments of increasing size from 0.008 to 300 grams in pressure equivalent
Measurement of pressure pain threshold on the operated hemithorax | Day 0 (day of surgery)
  An algogenic tip is applied with increasing pressure measured in grams checked on the monitor's digital screen. The subject will be educated to signal by applying a button (sound signal) when the required sensation (beginning pain) is reached.
Measurement of pressure pain threshold on the operated hemithorax | Visit 2 = 2 months after Day 0 (day of surgery)
  An algogenic tip is applied with increasing pressure measured in grams checked on the monitor's digital screen. The subject will be educated to signal by applying a button (sound signal) when the required sensation (beginning pain) is reached.
Measurement of pressure pain threshold on the unoperated hemithorax | Visit 2 = 2 months after Day 0 (day of surgery)
  An algogenic tip is applied with increasing pressure measured in grams checked on the monitor's digital screen. The subject will be educated to signal by applying a button (sound signal) when the required sensation (beginning pain) is reached.
Measurement of the vibration sensitivity threshold on the operated hemithorax | Day 0 (day of surgery)
  As soon as the subject perceives the vibration of the vibrameter, the value displayed on the digital panel will be noted. The operator will then increase the intensity a little then go back down. As soon as the patient no longer feels the vibration, the value displayed on the digital panel will be noted. The vibration perception value is obtained by calculating the average of the high and low values obtained.
Measurement of the vibration sensitivity threshold on the operated hemithorax | Visit 2 = 2 months after Day 0 (day of surgery)
  As soon as the subject perceives the vibration of the vibrameter, the value displayed on the digital panel will be noted. The operator will then increase the intensity a little then go back down. As soon as the patient no longer feels the vibration, the value displayed on the digital panel will be noted. The vibration perception value is obtained by calculating the average of the high and low values obtained.
Measurement of the vibration sensitivity threshold on the unoperated hemithorax | Visit 2 = 2 months after Day 0 (day of surgery)
  As soon as the subject perceives the vibration of the vibrameter, the value displayed on the digital panel will be noted. The operator will then increase the intensity a little then go back down. As soon as the patient no longer feels the vibration, the value displayed on the digital panel will be noted. The vibration perception value is obtained by calculating the average of the high and low values obtained.
Thermographic photo of the operated hemithorax | Day 0 (day of surgery)
  A camera coupled with a software makes it possible to identify changes in skin temperature. The region(s) clinically identified as pathological (neuropathic) will be identified beforehand by cutaneous tags (adhesive metallic controls that have been cooled beforehand).
Thermographic photo of the operated hemithorax | Visit 2 = 2 months after Day 0 (day of surgery)
  A camera coupled with a software makes it possible to identify changes in skin temperature. The region(s) clinically identified as pathological (neuropathic) will be identified beforehand by cutaneous tags (adhesive metallic controls that have been cooled beforehand).
Thermographic photo of the unoperated hemithorax | Visit 2 = 2 months after Day 0 (day of surgery)
  A camera coupled with a software makes it possible to identify changes in skin temperature. The region(s) clinically identified as pathological (neuropathic) will be identified beforehand by cutaneous tags (adhesive metallic controls that have been cooled beforehand).
Measurement of the conduction velocity in the operated hemithorax | Visit 2 = 2 months after Day 0 (day of surgery)
  A peripheral stimulation will be performed using a technique used in the intercostal region, and a cervical signal will be collected.
Measurement of the conduction velocity in the unoperated hemithorax | Visit 2 = 2 months after Day 0 (day of surgery)
  A peripheral stimulation will be performed using a technique used in the intercostal region, and a cervical signal will be collected.

SECONDARY OUTCOMES:
Total or partial pneumonectomy | Day 0 (day of surgery)
  Operative report
Operated side | Day 0 (day of surgery)
  Operative report
Number of drains | Day 0 (day of surgery)
  Operative report
Location of drains | Day 0 (day of surgery)
  Operative report
Importance of rib spacing | Day 0 (day of surgery)
  Operative report
Realization of perioperative epidural anesthesia | Day 0 (day of surgery)
  Operative report
Realization of thoracic paravertebral block | Day 0 (day of surgery)
  Operative report
Realization of intercostal block | Day 0 (day of surgery)
  Operative report
Response induced analgesia with topical lidocaine (in case of persistant pain) | Visit 2 = 2 months after Day 0 (day of surgery)
  Numeric scale of value (from 0 to 10)
Response induced analgesia to pregabalin (in case of persistent pain) | Visit 2 = 2 months after Day 0 (day of surgery)
  Numeric scale of value (from 0 to 10)

CONTACTS AND LOCATIONS:
Overall Officials: Christian DUALE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France